CLINICAL TRIAL: NCT03736226
Title: A Post-Approval, Single-Arm Study of the SYNERGYTM MONORAILTM Everolimus-Eluting Platinum Chromium Coronary Stent System in China
Brief Title: A Post-Approval, Single-Arm Study of the SYNERGY Stent System in China
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2424
Record Dates: First submitted 2018-07-30; First posted 2018-11-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: SYNERGYTM Stent System — no intervention design in the study

SUMMARY:
A prospective, observational, single-arm, open-label, multicenter, post-approval study. To compile real-world clinical outcomes data for the SYNERGYTM MONORAILTM Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGYTM Stent System) in real-world clinical practice in China.

DETAILED DESCRIPTION:
This prospective, open-label, multi-center study is designed to provide post-market surveillance information on the SYNERGY Stent System. The study will evaluate clinical outcomes of subjects receiving the SYNERGY™ stents over 5 years in a real world setting according to post approval requirements by China government.

ELIGIBILITY:
Inclusion Criteria:

* • Subject must be at least 18 years of age

  * Subject understands and provides written informed consent
  * Subject who is clinically indicated and will have an attempt of at least one SYNERGYTM stent OR Subject who is clinically indicated and was implanted with at least one SYNERGYTM stent
  * Subject is willing to comply with all protocol-required follow-up evaluation

Exclusion Criteria:

* Exclusion criteria are not required in this study which is an "all comers" study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "all comers" study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
MACE rate | 12 months
  endpoints will be assessed post stent implant

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China